CLINICAL TRIAL: NCT00746720
Title: Modulation of the Surgical Inflammatory Response by Etoricoxib: Peripheral Versus Central
Brief Title: Modulation of the Surgical Inflammatory Response by Etoricoxib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient recruitment difficulties
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: HELIOS Kliniken GmbH (Unknown); Rush University Medical Center (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02B2005; EudraCT No.: 2005-003854-80
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Pain; Osteoarthritis, Hip; Postoperative Pain
Keywords: hip replacement; osteoarthritis; etoricoxib; pain; cerebrospinal fluid; pharmacokinetics
MeSH Terms: conditions — Pain; Osteoarthritis, Hip; Pain, Postoperative; Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A, 1 (Experimental): Study part 1 (n = 8)
  Interventions: Drug: Etoricoxib 60 mg
- A, 2 (Placebo Comparator): Study part 1 (n = 4)
  Interventions: Drug: Placebo for Etoricoxib 60 mg
- B, 1 (Experimental): Study part 2 (n = 20)
  Interventions: Drug: Etoricoxib 60 mg
- B, 2 (Placebo Comparator): Study part 2 (n = 20)
  Interventions: Drug: Placebo for Etoricoxib 60 mg

INTERVENTIONS:
Drug: Etoricoxib 60 mg — film coated tablet 60 mg (orally), 120 mg (= 2 tablets a 60 mg) once daily, on day one post surgery
  Other Names: Arcoxia 60 mg; MK0663
  Arms: A, 1
Drug: Placebo for Etoricoxib 60 mg — film coated tablet (orally), two tablets once daily, on day one post surgery
  Other Names: Matching Placebo
  Arms: A, 2
Drug: Etoricoxib 60 mg — film coated tablet (orally), 120 mg (= 2 tablets a 60 mg) once daily, two hours before and 24 hours after surgery
  Other Names: Arcoxia 60 mg; MK0663
  Arms: B, 1
Drug: Placebo for Etoricoxib 60 mg — film coated tablet (orally), 2 tablets once daily, two hours before and 24 hours after surgery
  Other Names: Matching Placebo
  Arms: B, 2

SUMMARY:
The purpose of this study is to test the hypothesis that orally administered etoricoxib (COX-2) modulates prostaglandin and cytokine synthesis in the central nervous system (CNS) and in the periphery in surgical patients and thus reduces pain and suffering.

DETAILED DESCRIPTION:
This study will be a multiple centre, double-blind, placebo-controlled, randomized, parallel group study conducted in male and female adult patients undergoing elective primary single hip arthroplasty. In part 1 of the study 12 patients will be enrolled in the study and will be administrated 120 mg Etoricoxib or placebo orally on day one post surgery. The results from part 1 should help to adjust sampling time points (for blood, cerebrospinal fluid and hip drain fluid) if necessary. In part 2 of the study 40 patients will be enrolled and should receive 120 mg etoricoxib or placebo two hours before and 24 hours after surgery.

Primary end points will be the inflammatory mediators on peripheral and central levels. After surgical manipulation we expect increased mediators on both sides. It will be investigated if the medication could reduce the mediators compared to placebo and if the effect is related to pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing elective primary single hip arthroplasty
* Subject diagnosed with Osteoarthritis / arthrosis
* Subject has not taken non-steroidal anti-inflammatory drugs within 4 of their terminal half life times prior to enrollment
* Subject capable of understanding and cooperating with the requirements of the study

Exclusion Criteria:

* Patients with renal insufficiency (serum creatinine >1.5 mg/dl)
* Recent major trauma or systemic infection (within 3 months)
* Use of corticosteroid medication or chronic opioids (within 3 months)
* Any other condition likely to affect prostaglandin and cytokine levels
* Participation in another clinical study or receipt of an investigational drug within 30 days
* Hypersensitivity to any component of the etoricoxib and/or placebo tablets
* Uncontrolled hypertension defined as systolic blood pressure >140 mm Hg and diastolic pressure >90 mm Hg at rest after two repeated measurements
* Congestive heart failure (NYHA II-IV)
* Cerebrovascular disease
* Established ischemic heart disease (including patients who have recently undergone coronary artery bypass graft surgery or angioplasty)
* Patients with any kind or severity of cirrhosis of the liver or cholestasis or elevated liver function enzymes (ALT or AST 3 fold) as a sign of clinical significant liver malfunction (corresponds to any Child-Pugh-Score ≥5)
* Patients who have developed signs of asthma, acute rhinitis, nasal polyps, angioneurotic oedema or urticaria following the administration of aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Pregnancy and lactation
* Patients with active peptic ulcerations or active gastro-intestinal (GI) bleeding
* Inflammatory bowel disease
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or study site
* Any neurological syndrome or any other condition leading to contra-indication to spinal anesthesia

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that orally administered etoricoxib (COX-2 inhibitor) modulates prostaglandin and cytokine synthesis in the central nervous system (CNS) and in the periphery in surgical patients. | within 24 hours post dosing (study part 1) and within 48 hour post dosing (study part 2)

SECONDARY OUTCOMES:
To determine the CSF (cerebrospinal fluid), plasma and tissue pharmacokinetics of orally administered etoricoxib. | within 24 hours post dosing (study part 1) and within 48 hours post dosing (study part 2)
To correlate the prostaglandin and cytokine response to clinical outcome parameters after hip arthroplasty. | within 4 days post dosing (study part 1 and 2)
To assess the safety (via clinical laboratory tests and adverse events) of a single dose of 120 mg Etoricoxib for one day (Part1) or for two days (Part2) and placebo. | within 4 days post dosing (study part 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Brune, MD, PhD, Study Director — University of Erlangen-Nürnberg; Josef Zacher, MD, PhD, Principal Investigator — Helios Klinikum Berlin-Buch; Martin Fromm, MD, PhD, Principal Investigator — University of Erlangen-Nürnberg; Asokumar Buvanendran, MD, Principal Investigator — Rush University
Locations (1):
- HELIOS Klinikum Berlin, Berlin, Germany

REFERENCES:
- [Background] Buvanendran A, Kroin JS, Berger RA, Hallab NJ, Saha C, Negrescu C, Moric M, Caicedo MS, Tuman KJ. Upregulation of prostaglandin E2 and interleukins in the central nervous system and peripheral tissue during and after surgery in humans. Anesthesiology. 2006 Mar;104(3):403-10. doi: 10.1097/00000542-200603000-00005. PMID 16508385
- [Result] Renner B, Zacher J, Buvanendran A, Walter G, Strauss J, Brune K. Absorption and distribution of etoricoxib in plasma, CSF, and wound tissue in patients following hip surgery--a pilot study. Naunyn Schmiedebergs Arch Pharmacol. 2010 Feb;381(2):127-36. doi: 10.1007/s00210-009-0482-0. Epub 2010 Jan 6. PMID 20052461
- [Result] Renner B, Walter G, Strauss J, Fromm MF, Zacher J, Brune K. Preoperative administration of etoricoxib in patients undergoing hip replacement causes inhibition of inflammatory mediators and pain relief. Eur J Pain. 2012 Jul;16(6):838-48. doi: 10.1002/j.1532-2149.2011.00062.x. Epub 2011 Dec 19. PMID 22337568